CLINICAL TRIAL: NCT04399174
Title: 3DPD of the Placenta in Fetal Growth Restriction
Brief Title: Placental Vasculature for Prediction of Recurrent Fetal Growth Restriction
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, principal investigator, Benha University
Other Study IDs: khalid8
Record Dates: First submitted 2020-05-13; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Obstetric Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: US

SUMMARY:
: In this Prospective longitudinal observational study, two hundred pregnant women with singleton pregnancy from 11 up to 13 weeks with history of intrauterine growth restriction in a previous pregnancy underwent ultrasound assessment of gestational age , ultrasound assessment of uterine artery pulsatility index, placental volume by 3D ultrasound and placental vascularization by 3D power Doppler (3DPD).

DETAILED DESCRIPTION:
This Prospective longitudinal observational study was conducted at Benha University hospital starting from December 2016 to May 2019 after approval of faculty Research Ethics Board. Two hundred pregnant women with history of IUGR in previous pregnancy were recruited for the study after full explanation of the method, aim of work and obtaining consent. Inclusion criteria: singleton pregnancy from 11 up to 13 weeks. History of intrauterine growth restriction in previous pregnancy Exclusion criteria: Multiple pregnancies, Smoking women, and pre-existing medical disorders which may affect fetal growth e.g. hypertension, diabetes mellitus, thyroid dysfunction or renal impairment. Ultrasound evidence of congenital anomalies.

All women underwent ultrasound study which was performed by a member of ultra-sound unit (Volsun 730 pro V; G.E medical system), for assessment of: Gestational age confirmed by crown-rump length assessment, Uterine artery pulsatility index (angle of insonation is<50°, the sampling gate set at 2mm), 3D ultrasound assessment of Placental volume, 3DPD for assessment of placental vascularization. The examination was done with the patient in lithotomy position with slight left lateral tilting to avoid supine hypotension.

After visualization of the placental vasculature, 3D static power Doppler scanning was performed. After scanning the region of interest, placental volume was measured using the VOCAL rotational technique and VOCAL software (3D Sono View, GE Medical Systems, Milwaukee, WI, USA). After completing a full rotation, another analysis was performed using VOCAL Software (3D Sono View, GE Medical Systems, Milwaukee, WI, USA), which automatically calculates placental volume, vascularization index (VI), flow index (FI) and vascularization flow index(VFI). Low dose aspirin 75mg was described for all cases with the beginning of 2nd trimester.

All cases were having a second (between 20 to 24 weeks) and a third ultrasound assessment for exclusion of congenital malformation and assessment of fetal growth parameter and identification of IUGR cases (according to fetal growth curves). (Nicolaides KH et al., 2018). In order to avoid including healthy, yet constitutionally small for gestational age fetuses to the IUGR group, patients' data were included in the study only in cases of IUGR diagnosis confirmed after delivery.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy from 11 up to 13 weeks.
* History of intrauterine growth restriction in previous pregnancy

Exclusion Criteria: • Multiple pregnancies,

* Smoking women, and
* pre-existing medical disorders which may affect fetal growth e.g. hypertension, diabetes mellitus, thyroid dysfunction or renal impairment.
* Ultrasound evidence of congenital anomalies.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two hundred pregnant women with history of IUGR in previous pregnancy were recruited for the study after full explanation of the method, aim of work and obtaining consent.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
placental volume | 11-13 week
  Assessment of placental volume.
vascularization index (VI) | 11-13 week
  expressed as percentage, measures the number of colour voxels in the studied volume, representing the blood vessels within the tissue
uterine doppler | 11-13 week
  uterine artery pulsatility index
flow index (FI) | 11-13 week
  the average colour value of all colour voxels, representing average colour intensity.
vascularization flow index (VFI) | 11-13 week
  the average colour value of all grey and colour voxels, which represents both blood flow and vascularization

CONTACTS AND LOCATIONS:
Overall Officials: khalid salama, Principal Investigator — Benha University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ledee-Bataille N, Lapree-Delage G, Taupin JL, Dubanchet S, Frydman R, Chaouat G. Concentration of leukaemia inhibitory factor (LIF) in uterine flushing fluid is highly predictive of embryo implantation. Hum Reprod. 2002 Jan;17(1):213-8. doi: 10.1093/humrep/17.1.213. PMID 11756390
- See also: email of the principal investigator — http://dr,khalidsalama@gmail.com